CLINICAL TRIAL: NCT05704257
Title: Fetal Repair of Complex Gastroschisis: A Safety and Feasibility Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sundeep Keswani, Chief of Pediatric Surgery, Professor, Departments of Surgery, Pediatrics & OB/Gyn, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H-51929
Record Dates: First submitted 2023-01-03; First posted 2023-01-30 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Gastroschisis
Keywords: Gastroschisis; Abdominal Wall Defect
MeSH Terms: conditions — Gastroschisis | interventions — Fetoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- fetoscopic surgical repair (Experimental): Single arm study. All patients will receive the fetoscopic repair.
  Interventions: Device: fetoscopy

INTERVENTIONS:
Device: fetoscopy — The fetoscopic arm is described above. All patients will have a laparotomy, exteriorization of the uterus, and a fetoscopic repair of the gastroschisis.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and feasibility of fetal repair of complex gastroschisis (GS) via a fetoscopic surgical approach by assessing maternal, fetal, neonatal, and infant outcomes in a cohort of 10 patients. The hypothesis is that in utero repair of GS will reduce postnatal mortality and morbidity in complex GS infants with minimal maternal and fetal risk.

DETAILED DESCRIPTION:
Gastroschisis is a congenital abdominal wall defect by which the intestinal structures eviscerate from the abdomen, with a current prevalence of 4.9 per 10,000 pregnancies in the United States. Not only is it the most common abdominal wall defect, but the incidence of GS has increased by nearly 30% in the US (Jones et al., 2016) and 25 % in Europe (EUROCAT, 2021) between 2006 and 2012 for reasons that are still unknown. Two subtypes of the disease have been identified - simple and complex GS. Simple GS presents as an otherwise healthy bowel that may have an inflammatory peel over the bowel surface. By contrast, complex GS is characterized by serious bowel complications, such as bowel volvulus, atresia, stenosis, necrosis, and perforation.

Participants will be offered the minimally invasive in-utero repair technique as an alternative to the traditional standard postnatal GS surgical repair. During surgery, the mother's uterus is opened using the standard laparotomy approach that we currently use in our open fetal surgeries and fetoscopic spina bifida repair through an exteriorized uterus, and then fetal surgeons repair the fetus' defect. The uterus is closed, and the pregnancy continues. When babies are treated in this way, they may be less likely to be born with their intestines coming out of their belly and if this is the case, they may be less likely to have other problems that occur with gastroschisis because the intestines are not covered.

All participants will be closely followed with ultrasound and consultation after the surgery. Delivery will be scheduled at Texas Children's Hospital, and the infants will be followed for 12 months by our research team.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women - maternal age 18 years or older and capable of consenting for her own participation in this study
2. Singleton pregnancy
3. Sonographic evidence of gastroschisis (exteriorization of bowel content outside the fetal abdominal cavity into the amniotic cavity)
4. Intraabdominal bowel dilation ≥ 8 mm at 20-24 weeks GA reviewed by prenatal ultrasound
5. Absence of significant associated anomalies* diagnosed on prenatal ultrasound or MRI
6. Gestational age at the time of the procedure will be between 20 0/7 weeks and 25 6/7 weeks
7. Absence of chromosomal and clinically significant abnormalities, i.e., normal karyotype and/or normal chromosomal microarray (CMA) by invasive testing (amniocentesis or Chorionic Villus Sampling (CVS)). If there is a balanced translocation with normal CMA with no other anomalies the candidate can be included. Results by fluorescence in situ hybridization (FISH) will be accepted, if the candidate's gestation age is ≥ 22 0/7 weeks. Patients declining invasive testing will be excluded
8. The family has considered and declined the option of termination of the pregnancy at less than 24 weeks and of standard postnatal treatment
9. The family meets psychosocial criteria (sufficient social support, ability to understand the requirements of the study)
10. Parental/guardian permission (informed consent) for follow up of the child after birth

    * Significant associated anomalies are defined as such anomalies that would, in and of themselves, be life limiting or life threatening. A minor anomaly, such as a small VSD or ASD not deemed to be life limiting or threatening, or a cleft lip or other such anomaly, unless part of a genetic syndrome, will not disqualify the patient.

Exclusion Criteria:

1. Significant fetal anomaly unrelated to gastroschisis
2. Evidence of bowel perforation (presence of intraabdominal bowel calcification on ultrasonography)
3. Increased risk for preterm labor including short cervical length (≤ 2.0 cm), history of incompetent cervix with or without cerclage, and previous preterm birth in a singleton pregnancy (other than a patient delivered for a non-repeating medical or surgical indication)
4. Placental abnormalities (previa, abruption, accreta) known at time of enrollment
5. Pre-pregnancy body-mass index (BMI) ≥40
6. Contraindications to surgery including previous hysterotomy (whether from a previous classical cesarean, uterine anomaly such as an arcuate or bicornuate uterus, major myomectomy resection, or previous fetal surgery) in active uterine segment
7. Technical limitations precluding fetoscopic surgery, such as extensive uterine fibroids, fetal membrane separation, or uterine anomalies
8. Maternal-fetal Rh alloimmunization, Kell sensitization, or neonatal alloimmune thrombocytopenia affecting the current pregnancy.
9. Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment
10. Maternal medical condition that is a contraindication to surgery or general anesthesia
11. Low amniotic fluid volume (Amniotic Fluid Index less than 6 cm) if deemed to be due to fetal anomaly, poor placental perfusion or function, or membrane rupture. Low amniotic fluid volume that responds to maternal hydration is not an exclusion criterion
12. Patient does not have a support person (i.e., spouse, partner, or mother) available to support her for the duration of the pregnancy
13. Inability to comply with the travel and follow-up requirements of the trial
14. Patient scores as severely depressed on the Edinburgh Postnatal Depression Scale (EPDS)
15. Patients that are enrolled or have been enrolled in any another intervention study that affects the mother or fetus
16. Maternal hypersensitivity to any of the entities associated w/ AlloDerm™. The use of AlloDerm™ Regenerative Tissue Matrix distributed by Allergan Aesthetics is contraindicated for patients sensitive to any of the antibiotics listed on the AlloDerm package, i.e., Gentamycin, Cefoxitin, Lincomycin, Polymyxin B and Vancomycin or Polysorbate 20

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Successful Repair of Complex Gastroschisis | At end of surgical repair
  Success of primary skin closure after complete bowel reduction.

SECONDARY OUTCOMES:
Intrauterine Fetal Death (IUFD) | At delivery
  Demise of fetus while still in the womb
Preterm Birth | At delivery
  Number of patients that deliver at < 37 weeks gestation
Time to initiation of enteral feeds (days) | At hospital discharge, an average of 1.5 months
  The number of days until initiation of enteral feeding
Time on total parenteral nutrition (TPN) (days) | At hospital discharge, an average of 1.5 months
  The number of days on total parenteral nutrition (TPN)
Necrotizing Enterocolitis | At hospital discharge, an average of 1.5 months
  As measured by presence in medical record
Short Bowel Syndrome | At hospital discharge, an average of 1.5 months
  As measured by presence in medical record
Length of Hospital Stay | At the time of discharge from the NICU, an average of 1.5 months
  Length of stay in the hospital measured in days
Intracranial hemorrhage | During first month of life
  Measured as presence in neonate during first month by MRI and/or ultrasound.
Retinopathy of Prematurity | At the time of discharge from the NICU, an average of 1.5 months
  Postnatal grade classification presence of grade III or higher using standardized system (yes/no)
Respiratory Distress Syndrome | At the time of discharge from the NICU, an average of 1.5 months
  As measured by presence in medical record
Bronchopulmonary Dysplasia | At the time of discharge from the NICU, an average of 1.5 months
  As measured by presence in medical record
Need for Gastroschisis related surgery | 12 months of age
  As measured by presence in medical record ≤12 months
Small Bowel Obstruction | 12 months of age
  As measured by presence in medical record ≤12 months
Central Line Associated Bloodstream Infection (CLABSI) | 12 months of age
  As measured by presence in medical record ≤12 months
Neuro-developmental Outcome at 12 months | 12 months of age
  As measured by the Capute Scales at 12 months
Survival at 12 months | 12 months of age
  Number of patients alive at 12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Sundeep Keswani, MD, Principal Investigator — Baylor College of Medicine and Texas Children's Hospital
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States